CLINICAL TRIAL: NCT03484546
Title: Optimum Menstrual Cycle Time for Endometrioma Excision
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Turgut Aydın, Assistant Professor, Acibadem University
Other Study IDs: AcibademGynecology
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Endometriosis; Endometrioma
Keywords: ovarian reserve; endometriosis; endometrioma
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- folicular: Women who will undergo endometrioma cystectomy in her follicular phase of menstrual period.
  Interventions: Procedure: laparoscopic endometrioma cyst excision
- ovulatory: Women who will undergo endometrioma cystectomy in her ovulatory phase (12-14th day of mestrual period cycle for women regular period) of menstrual cycle.
  Interventions: Procedure: laparoscopic endometrioma cyst excision
- luteal: Women who will undergo endometrioma cystectomy in her luteal phase of menstrual period.
  Interventions: Procedure: laparoscopic endometrioma cyst excision

INTERVENTIONS:
Procedure: laparoscopic endometrioma cyst excision — laparoscopic resection of ovarian endometrioma

SUMMARY:
This study evaluates the optimum day of menstrual period for the excision of endometriomas to minimize the damage of surgery to normal ovarian tissue. Patients will be grouped as follicular, ovulatory and luteal according to menstrual days. Ovarian damage will be evaluated with both pathologic examination and anti-mullerian hormone levels before and after the surgery.

DETAILED DESCRIPTION:
Endometriosis is a common gynecologic disease seen in about 10% of women in reproductive age. The most common site of endometriosis is overt. Cystic formation of ovarian endometriosis is called endometrioma (chocolate cyst). Definitive treatment of endometriomas is excision by laparoscopy. The disadvantage of this surgery is the removal of some of the normal ovarian follicles within cystectomy material. This procedure can damage the ovarian reserves with the treatment of endometriomas, which are already the cause of infertility, and lead to the conditions such as infertility or early menopause. It has been understood that the ovarian reserves of the patients who underwent endometrioma cystectomy with the decrease of the Anti-Mullerian Hormone values, which is an over reserve parameter.

ELIGIBILITY:
Inclusion Criteria:

* 4 to 10 cm unilateral ovarian endometrioma
* having clinically indication of laparoscopic ovarian endometrioma excision

Exclusion Criteria:

* prior gynecologic surgery
* prior abdominal surgery
* additional operation in the same session
* having the diagnosis of premature ovarian failure or ovarian insufficiency
* having any diagnosis of malignancy
* having diagnosis of a non-gynecologic chronicle disease

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who admitted to out-patient clinic between the ages of 18-40 years,had 4-10cm ovarian unilateral endometrioma and had an indication of laparoscopic ovarian endometrioma excision.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Determination of ovarian follicle damage via histological examination | 5 days after the surgery
  Histologic evaluation of the cystectomy excision material for health ovarian follicles
Change of anti-mullerian hormone level 6 months after surgery | 6 months
  Comparison of pre-operative and 6 months after surgery of anti-mullerian hormone levels

CONTACTS AND LOCATIONS:
Overall Officials: Ozguc Takmaz, Principal Investigator — Acibadem MAA University Maslak Hospital
Locations (3):
- Turkey (Türkiye) (3):
  - Acibadem Fulya Hospital, Istanbul
  - Acibadem MAA University Atakent Hospital, Istanbul
  - Acibadem MAA University Maslak Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will be decided during the study process.

REFERENCES:
- [Derived] Takmaz O, Asoglu MR, Ceyhan M, Unsal G, Gungor M. Comparing ovarian reserve parameters after laparoscopic endometrioma resection in the follicular vs. luteal phase: a prospective cohort study. Front Med (Lausanne). 2024 Oct 15;11:1469858. doi: 10.3389/fmed.2024.1469858. eCollection 2024. PMID 39473503